CLINICAL TRIAL: NCT02899910
Title: Nutrition and Exercise Study to Understand Metabolic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Gurjeet Birdee, Principle Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Vanderbilt University
Record Dates: First submitted 2016-09-06; First posted 2016-09-14 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Metabolic Syndrome; Obesity; Insulin Resistance
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Insulin Resistance | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Yoga with health education (Experimental): 12 week yoga program coupled to standardized health education for weight loss
  Interventions: Behavioral: Health education; Behavioral: Yoga
- Health education (Active Comparator): Standardized health education for weight loss
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Health education — Education on lifestyle changes for treatment of metabolic syndrome
Behavioral: Yoga — Training in the practice of yoga for treatment of metabolic syndrome
  Arms: Yoga with health education

SUMMARY:
The purpose of this study is to measure the metabolic and behavioral effects of a 12-week yoga program coupled to health education (HED) compared to HED alone.

DETAILED DESCRIPTION:
The purpose of this study is to measure the metabolic and behavioral effects of a 12-week yoga program coupled to health education (HED) compared to HED alone. In a randomized clinical trial of 90 patients (45 patients per arm), investigators will measure the effects of the two interventions on IR, HTN, dysplidemia, and body composition (See Figure 1. Study Diagram). Subjects will be scheduled for outcome assessment at baseline, 12 weeks, and 24 weeks. In addition, investigators will collect data at baseline and 12 weeks on self-efficacy, stress, mindfulness, and mood. As a sub-study to the randomized controlled trial, investigators will measure the aerobic intensity of the yoga to estimate the dose of physical exercise provided by the yoga (n=10).

Subjects willing and eligible to participate in the RCT will receive written consent. Consented subjects will be randomized to either 12 weeks of yoga with HED versus HED alone. Subjects randomized to yoga will receive 30 to 45 minutes of weekly yoga instruction, followed by 30 to 45 minutes of HED. Subjects will receive written instructions for home yoga practice and lifestyle changes based on HED. Subjects randomized to HED alone will receive a weekly standardized HED curriculum which will be attention and time matched to the yoga with HED arm.

ELIGIBILITY:
Inclusion Criteria:

* Elevated waist circumference (Men greater than 102cm; women greater than 88cm)
* Impaired fasting glucose (100-125 mg/dl)
* Elevated blood pressure (systolic ≥130 and/or diastolic ≥ 85)
* Dyslipidemia (triglycerides ≥150 and/or HDL≤ 40 for men; 50 for women)
* Age ≥ 18
* English speaking

Exclusion Criteria:

* Currently taking blood pressure medications, oral diabetic medication or insulin, or lipid medication
* Systolic blood pressure ≥160 and/or diastolic ≥100
* Unstable cardiac disease e.g. angina, life threatening arrhythmia
* Lung disease requiring oxygen supplementation at rest or with ambulation
* History of dementia or cognitive impairment
* Uncontrolled psychiatric disorders, such as major depression or psychosis
* Current participation in a mind-body practice/program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in insulin resistance | Baseline, 12 weeks, and 24 weeks

SECONDARY OUTCOMES:
Change in hypertension | Baseline, 12, and 24 weeks
  Blood pressure
Change in dyslipidemia | Baseline, 12, and 24 weeks
  Fasting lipids
Change in body composition | Baseline, 12, and 24 weeks
  Waist circumference and bioelectrical impedance
Change in diet | Baseline, 12, and 24 weeks
  Dietary intake assessed with Block Brief 200 Food Frequency
Change in physical activity measured with accelerometers | Baseline, 12, and 24 weeks
  Assessed with accelerometers
Change in self-efficacy | Baseline and 12 weeks
  Perceived Health Competence Scale
Change in stress | Baseline and 12 weeks
  Perceived Stress Scale-10
Change in quality of life | Baseline and 12 weeks
  SF-36
Change in mindfulness | Baseline and 12 weeks
  Mindful Attention and Awareness Scale
Change in affect measured through questionnaire Profile of Mood States | Baseline and 12 weeks
  Profile of Mood States

CONTACTS AND LOCATIONS:
Overall Officials: Gurjeet Birdee, MD, Principal Investigator — Vanderbilt University Medical Center

IPD SHARING:
Plan to Share IPD: No